CLINICAL TRIAL: NCT03113513
Title: Randomized Trial of Sacrospinous Ligament Fixation Versus McCall Culdoplasty in Women Undergoing Vaginal Hysterectomy and Repairs for Prolapse
Brief Title: Comparison of Two Apical Repair Methods in Women Undergoing Repairs for Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V4 31.01.2016
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Pelvic Organ Prolapse; Surgery; Quality of Life; Complication
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: The study is designed as a RCT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McCall culdoplasty (Active Comparator): The McCall culdoplasty will be performed in a modified version as described by McCall in 1957. Specifically, two long acting bioresorbable sutures are put through the specific anatomic landmarks.
  Interventions: Procedure: fixation of the vaginal apex
- Sacrospinous ligament fixation (Active Comparator): The SLF technique will be performed as described by Richter et al (Amreich, 1951). Two long acting bioresorbable sutures are passed through the right sacrospinous ligament and then fixed to the vaginal cuff.
  Interventions: Procedure: fixation of the vaginal apex

INTERVENTIONS:
Procedure: fixation of the vaginal apex — In the course of vaginal hysterectomy the vaginal cuff is either fixed to the sacrospinous ligament or to the uterosacral ligament.

SUMMARY:
To date no study has determined prospectively which technique is superior to prevent recurrent Pelvic Organ Prolapse (POP) after vaginal hysterectomy- a major unmet clinical need. The aim of the study is to determine objective anatomical recurrent prolapse after Sacrospinous Ligament Fixation (SLF) vs McCall.

DETAILED DESCRIPTION:
The aim of the study is to determine objective anatomical recurrent prolapse after SLF vs McCall. The study is designed as a Randomized Controlled Trial (RCT). Primary study endpoint will be at 12 months, secondary study endpoint at 24 months. The following parameters will be evaluated after one year: anatomical outcome, Quality of Life (QoL), sexual health, reoperations, and complications.

ELIGIBILITY:
Inclusion Criteria:

* declined/ failed conservative treatment for POP
* planned vaginal hysterectomy with anterior/posterior colporrhaphy as indicated
* any symptomatic POP or stage II prolapse in any compartment
* at least stage I prolapse in the apical department
* women between 35 and 80 years of age
* good German language skills
* any concomitant prolapse surgery (anterior, posterior vaginal repair, suburethral tapes) as indicated
* concomitant salpingo-oophorectomy if indicated

Exclusion Criteria:

* Unwillingness to participate
* Neurological disorders
* Previous hysterectomy
* Desire to have children
* Connective tissue disorders (i.e. Ehlers-Danlos syndrome, Marfan syndrome)

Ages: 35 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — only women are included into the study
Enrollment: 312 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with stage 2 or higher on the Pelvic Organ Prolapse Quantification System (POP-Q). | 12 months after surgery
  POP-Q stage 2 or higher means any point of the POP-Q system being -1 related to the hymen or below

SECONDARY OUTCOMES:
Subjective cure | 12 months after surgery
  determined by the Patient Global Impression of Improvement (PGII) index
Quality of life as determined by a questionnaire | 12 months after surgery
  The Kings Health Questionnaire was validated in women with stress urinary incontinence and assesses the impact of incontinence on quality of life. The eight subscales ("domains") scored between 0 (best) and 100 (worst). The Symptom Severity scale is scored from 0 (best) to 30 (worst); lower scores indicate better QoL. Success in terms of the study is defined as 10 points improvement on the total Kings Health Questionnaire score.
Sexual health | 12 months after surgery
  The Pelvic Organ Prolapse Incontinence Sexual Questionnaire is a 20 item questionnaire and is the primary measure used to assess sexual function in women with urinary incontinence and prolapse. Mean subscale scores are calculated by summing the valid responses to items in the subscale and then divided by the number of items with valid responses. The higher the subscores, the worse the outcome.
Reoperation rate | 12 months after surgery
  Number of patients with any reoperations for POP

CONTACTS AND LOCATIONS:
Locations (1):
- MUGRAZ, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No
The sponsor has access to all study relevant data. In the specific centers only authorized study personnel has access to the data.

REFERENCES:
- [Background] Colombo M, Milani R. Sacrospinous ligament fixation and modified McCall culdoplasty during vaginal hysterectomy for advanced uterovaginal prolapse. Am J Obstet Gynecol. 1998 Jul;179(1):13-20. doi: 10.1016/s0002-9378(98)70245-5. PMID 9704759